CLINICAL TRIAL: NCT07084818
Title: Enabling Self-Care for Pessary Users in Rural Setting
Acronym: ESCAPE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, Kris.Strohbehn, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02003005
Record Dates: First submitted 2025-07-23; First posted 2025-07-25 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pessary; Pelvic Organ Prolapse; Self-Care; Rural Care
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Intervention group will be subjects trying new collapsible pessary and providing self-care of their pessary. Control group will be subjects continuing with their current pessary and office-based care of their pessary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Self-Care (Experimental): Subjects who switch to new, collapsible pessary and convert to self-management for care of their pelvic organ prolapse.
  Interventions: Device: Reia System pessary self-care management
- Office-Care (Active Comparator): Subjects who continue office-based pessary care of their pelvic organ prolapse with visits every 3-6 months annually.
  Interventions: Device: Standard pessary office-based management

INTERVENTIONS:
Device: Reia System pessary self-care management — The Reia-System pessary is an FDA-cleared device to manage pelvic organ prolapse which is collapsible and intended to be more easily removed, with less discomfort.
  Other Names: collapsible pessary
  Arms: Self-Care
Device: Standard pessary office-based management — These subjects will continue with the current pessary they are using to manage their prolapse, with office-based care.
  Other Names: Ring pessary, Gellhorn pessary, donut pessary, cube pessary
  Arms: Office-Care

SUMMARY:
This study is to see if a using new collapsible pessary (Reia pessary) for treatment of pelvic organ prolapse will allow patients to care for their prolapse on their own, rather than having to come to be seen by a provider in the office regularly (2-4 times per year) to manage the pessary. Enrollment in the study will be offered to current patients who have regular office visits to care for their pessary.

DETAILED DESCRIPTION:
This is a prospective interventional trial for patients with at least stage 2 pelvic organ prolapse (POP), who are currently managing their POP with office-based care using a pessary. The study will be conducted at two institutions, Dartmouth-Hitchcock and Pennsylvania State University. The intervention will be to convert willing patients from office-based care to self-care, using a new, collapsible (Reia) pessary in patients. The primary outcome will be a visual analog score (VAS) regarding their current satisfaction with their treatment and management of POP. Secondary outcomes will include questionnaires on impact, travel for care and self-care. The comparison group will be patients who decline to try the new pessary but agree to questionnaires regarding their current office-based care for pessary management.

ELIGIBILITY:
Inclusion Criteria:

* Women currently using office-based pessary management of at least stage 2 POP will be recruited:
* English-speaking natal females 18 years or older
* Stage II-IV POP desiring continued pessary management.
* Primary indication for pessary management is treatment of POP

Exclusion Criteria:

* Primary indication for pessary is for management of stress urinary incontinence
* Vesicovaginal fistula or rectovaginal fistula
* Vaginal, rectal or bladder malignancy
* Genitourinary infection requiring treatment*
* Ongoing treatment for vaginal infections (e.g., chronic bacterial vaginosis)*
* Inflammatory bowel disease (Crohn's or ulcerative colitis)
* Pelvic or anorectal chronic pain
* Pelvic floor surgery within the past 6 months or planning to undergo pelvic floor surgery
* Congenital malformation of the bladder, rectum or vagina
* The following special populations will be excluded:

Adults unable to consent Individuals who are not yet adults (infants, children, teenagers) Pregnant women (or planning pregnancy in the next 6 months) (women of childbearing age will be verbally queried and offered pregnancy testing if uncertain) Prisoners

*Patients with acute vaginal infections will be eligible for enrollment 2 weeks after completing treatment and have resolution of symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants are eligible females with pelvic organ prolapse (POP) who are currently managing with a pessary. POP is a gender-specific condition only affecting females.
Enrollment: 120 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score (VAS): satisfaction of prolapse management. | Baseline, 3 months, 6 months
  Patient reported Visual Analogue Score for (0-100mm) for satisfaction of prolapse management.

SECONDARY OUTCOMES:
modified Patient Experience with Treatment and Self-Management (mPETS) Questionnaire | Baseline, 6 months
  modified Patient Experience with Treatment and Self-Management Questionnaire. This is a 41-item questionnaire that is validated for patient experience with treatment and self-management of diseases as a measure of treatment burden. The questionnaire has been shortened from the original 48-item questionnaire in the original study by Eton et al and it has been slightly modified to address how prolapse and pessary care impacts treatment burden. Minimum value = 41, Maximum value = 205. Higher PETS scores are associated with greater treatment burden, with more distress, less satisfaction with medications, lower self-efficacy, worse physical and mental health, and lower convenience of healthcare.
Patient Experience with Pessary Treatment and Self-Management (PEPS) Questionnaire | Baseline, 6 months
  Patient Experience with Pessary Treatment and Self-Management Questionnaire. This is a non-validated 11-item questionnaire that is focused on factual information regarding patient's care of their prolapse, including how long they have used a pessary, if they have cared for it themselves, how far they travel for care, how often they have their pessary checked by a practitioner. There are a few individual scaled questions with Likert responses, regarding discomfort of pessary removal and reinsertion (0-4, with the highest score being the worst outcome, "very uncomfortable"); bother of care for the pessary (0-5, the highest score being the worst outcome, "very bothersome"); interest in taking care of the pessary (0-5, the highest score being the worst outcome, "not interested at all". There is one visual analogue score (minimum 0, maximum 10) on how bothersome it is to have to travel for office care several times per year.
Pelvic Floor Impact Questionnaire - 7 (PFIQ-7) | Baseline, 6 months
  Pelvic Floor Impact Questionnaire - 7. This is a validated 7-item questionnaire that assesses treatment on pelvic floor impact for urinary symptoms, prolapse symptoms and colorectal symptoms. Each of the seven questions for each symptom category (bladder, prolapse, rectal) has a scale of 0-3, with higher scores being worse. The total PFIQ-7 score range is 0-300, with the higher score being worse. It has been used in many studies on prolapse, including preliminary studies on the Reia pessary.
Pessary Sexual Questionnaire | Baseline, 6 months
  This is a non-validated 8-item questionnaire on sexual activity for subjects and whether the pessary impacts ability to be sexually active. Most questions are informational yes/no responses. The last question is a Likert scale [0-3] regarding how much the current pessary interferes with being able to be sexually active, with 3 being worse, "interferes a lot".
Patient Global Impression of Improvement (PGI-I) | 3 months, 6 months
  Patient Global Impression of Improvement: Validated one-item questionnaire (Likert scale, 1-7); The highest score is a worse outcome.
Patient Global Impression of Severity (PGI-S) | Baseline, 3 months, 6 months
  Patient Global Impression of Severity: Validated one-item assessment of severity of prolapse condition (Likert scale, 1-4). The highest score is a worse outcome.
Patient Global Symptoms Rating Scale (PGSC) | Baseline, 3 months, 6 months
  Patient Global Symptoms Rating Scale (PGSC): Non-validated one-item questionnaire of treatment and adequacy of control of symptoms (Likert scale, 1-5); The highest score is a better outcome.
Number of subjects with at least one adverse event | 0-6 months
  Adverse events will be collected, including discharge, bleeding, pain during the course of the study in both the intervention group and the continued office-based care group. There is not a maximum number of adverse events but a The highest number is a worse outcome.
Log of pessary self-care events | 0-6 months
  Patients who decide to learn self-management of their pessary will record the number of times they remove and reinsert the pessary.

CONTACTS AND LOCATIONS:
Overall Officials: Kris Strohbehn, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strohbehn K, Wadensweiler PM, Richter HE, Grimes CL, Rardin CR, Rosenblatt PL, Toglia MR, Siddiqui G, Hanissian P. Effectiveness and safety of a novel, collapsible pessary for management of pelvic organ prolapse. Am J Obstet Gynecol. 2024 Aug;231(2):271.e1-271.e10. doi: 10.1016/j.ajog.2024.05.009. Epub 2024 May 16. PMID 38761837
- [Background] Strohbehn K, Wadensweiler P, Hanissian P. A novel, collapsible, space-occupying pessary for the treatment of pelvic organ prolapse. Int Urogynecol J. 2023 Jan;34(1):317-319. doi: 10.1007/s00192-022-05415-y. Epub 2022 Dec 3. No abstract available. PMID 36462059
- [Background] Eton DT, Yost KJ, Lai JS, Ridgeway JL, Egginton JS, Rosedahl JK, Linzer M, Boehm DH, Thakur A, Poplau S, Odell L, Montori VM, May CR, Anderson RT. Development and validation of the Patient Experience with Treatment and Self-management (PETS): a patient-reported measure of treatment burden. Qual Life Res. 2017 Feb;26(2):489-503. doi: 10.1007/s11136-016-1397-0. Epub 2016 Aug 26. PMID 27566732
- [Background] Chen X, Orom H, Hay JL, Waters EA, Schofield E, Li Y, Kiviniemi MT. Differences in Rural and Urban Health Information Access and Use. J Rural Health. 2019 Jun;35(3):405-417. doi: 10.1111/jrh.12335. Epub 2018 Nov 16. PMID 30444935
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Srikrishna S, Robinson D, Cardozo L. Validation of the Patient Global Impression of Improvement (PGI-I) for urogenital prolapse. Int Urogynecol J. 2010 May;21(5):523-8. doi: 10.1007/s00192-009-1069-5. Epub 2009 Dec 15. PMID 20013110
- [Background] Kearney R, Brown C. Self-management of vaginal pessaries for pelvic organ prolapse. BMJ Qual Improv Rep. 2014 Oct 21;3(1):u206180.w2533. doi: 10.1136/bmjquality.u206180.w2533. eCollection 2014. PMID 27493737
- [Background] Dwyer L, Rajai A, Dowding D, Kearney R. Understanding Factors That Affect Willingness to Self-Manage a Pessary for Pelvic Organ Prolapse: A Questionnaire-Based Cross-Sectional Study of Pessary-Using Women in the UK. Int Urogynecol J. 2024 Aug;35(8):1627-1634. doi: 10.1007/s00192-024-05840-1. Epub 2024 Jul 2. PMID 38953998
- [Background] Sung VW, Jeppson P, Madsen A. Nonoperative Management of Pelvic Organ Prolapse. Obstet Gynecol. 2023 Apr 1;141(4):724-736. doi: 10.1097/AOG.0000000000005121. Epub 2023 Mar 9. PMID 36897185